CLINICAL TRIAL: NCT01074489
Title: Challenging the Gold Standard: A Pilot Study Comparing CGMS and Capillary Glucose Monitors Versus 3 Hour GTT to Diagnose Gestational Diabetes Mellitus
Brief Title: Challenging the Gold Standard: Pilot Study Comparing Continuous Glucose Monitoring System (CGMS), Capillary Glucose Monitors and 3 Hour Glucose Tolerance Test (GTT) to Diagnose Gestational Diabetes Mellitus (GDM)
Status: Completed | Type: Observational
Sponsor: University of Cincinnati (Other)
Responsible Party: Principal Investigator, Ronald Jaekle, Professor, University of Cincinnati
Other Study IDs: GDM Gold 1
Record Dates: First submitted 2010-02-22; First posted 2010-02-24 (Estimated); Last update posted 2015-08-25 (Estimated); Status verified 2015-08

CONDITIONS: Diabetes, Gestational
Keywords: GDM; Gestational Diabetes; GTT; CGMS
MeSH Terms: conditions — Diabetes, Gestational

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this research study is to compare 3 methods of measuring blood glucose (blood sugar) levels to see if the finger-stick method or the continuous glucose monitoring system is better than or as good as the 3 hour glucose tolerance test (GTT) for the diagnosis of gestational diabetes.

DETAILED DESCRIPTION:
The rate of gestational diabetes and fetal macrosomia is increasing. Moreover, it appears that many macrosomic infants are born to non-diabetic mothers. However, this presents the question of whether our current accepted means of diagnosis is reflecting the true prevalence of GDM. The 3-hour GTT measures glycemic control over a limited period of time. A more prolonged period of monitoring makes more physiologic sense, as it would paint a picture of a patient's overall trend before a diagnosis can be confirmed or excluded. Given the ability of the CGMS and capillary glucose monitor to follow glycemic trends over an extended time period, these methods may prove more effective at identifying patients with abnormal glucose tolerance. As these modalities test the patients in their native environments, the effect of dietary changes prior to the testing period may be minimized, potentially providing an more accurate assessment of abnormal glucose utilization. Furthermore, both modalities should be more cost-effective than the 3- hour GTT.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant patients seen in the Center for Women's Health at University Hospital in Cincinnati, Ohio between 24-28 weeks gestation
* One hour 50-g Glucose Challenge Test (GCT) value greater than 130 mg/dL.

Exclusion Criteria:

* Patients with known diabetes mellitus
* Patients receiving steroids or oral terbutaline therapy
* Patients entering prenatal care later than 20 weeks gestation

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Pregnant women between 18 & 50 years old who are having a 3 hour GTT as directed by their doctor
Sampling Method: Non-Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2010-02; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Blood glucose levels | Over 1 week

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Jaekle, MD, Principal Investigator — University of Cincinnati
Locations (1):
- University of Cincinnati, Cincinnati, Ohio, United States

REFERENCES:
- [Background] Harlass FE, Brady K, Read JA. Reproducibility of the oral glucose tolerance test in pregnancy. Am J Obstet Gynecol. 1991 Feb;164(2):564-8. doi: 10.1016/s0002-9378(11)80021-9. PMID 1992702
- [Background] Melki V, Ayon F, Fernandez M, Hanaire-Broutin H. Value and limitations of the Continuous Glucose Monitoring System in the management of type 1 diabetes. Diabetes Metab. 2006 Apr;32(2):123-9. doi: 10.1016/s1262-3636(07)70258-6. PMID 16735960
- [Background] Rivers SM, Kane MP, Bakst G, Busch RS, Hamilton RA. Precision and accuracy of two blood glucose meters: FreeStyle Flash versus One Touch Ultra. Am J Health Syst Pharm. 2006 Aug 1;63(15):1411-6. doi: 10.2146/ajhp050473. PMID 16849704